CLINICAL TRIAL: NCT03462550
Title: A Randomized Study Comparing the Laryngeal Mask Airway Supreme With the Laryngeal Mask Airway Protector In the Ambulatory Surgery Unit
Brief Title: A Study Comparing the Laryngeal Mask Airway Supreme With the Laryngeal Mask Airway Protector In the Ambulatory Surgery Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/2017/0117
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Airway Complication of Anesthesia
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LMA Supreme (Active Comparator)
  Interventions: Device: Laryngeal mask
- LMA Protector (Experimental)
  Interventions: Device: Laryngeal mask

INTERVENTIONS:
Device: Laryngeal mask — LMA insertion

SUMMARY:
The Laryngeal Mask Airway is a supraglottic airway device that has been used in anesthesia for decades. Now the third generation (LMA Supreme) is commonly used. Recently the LMA Protector is manufactured.

The primary hypothesis of this study is: the oropharyngeal leak pressure of the LMA Protector is 5 cmH2O higher than the oropharyngeal leak pressure of the LMA Supreme. Secondary outcome measures are: ease of insertion, fibreoptic position, ease of gastric tube placement.

Differences between LMA Supreme and LMA Protector are: the LMA protector has a dual gastric drainage channel, LMA supreme one. For LMA protector, airway tube and cuff are 100% silicone, in LMA supreme the cuff is polivinylchloride. Silicone cuffs have shown to reduce risk of sore throat and achieve higher seal pressures. There are no aperture bars in the LMA protector (2 in LMA supreme). The tube of LMA protector is more flexible. An integrated cuff pressure indicator for single use airway management devices that enables continuous cuff pressure monitoring only in the LMA protector.

DETAILED DESCRIPTION:
1. Outpatients planned for elective minor surgery, routinely done with LMA, will be asked to participate in the study.
2. The patient is preoxygenated for 3 min. Anaesthesia is induced with 0.15 mcg/kg sufentanil and 1 - 4 mg/kg propofol. Routine monitoring is used together with BIS-monitoring. No neuromuscular relaxing agent is used. Patients lungs will be ventilated with a face mask for 3 min and then the LMA will be inserted while the neck of the patient is flexed, the head extended. LMA cuff is completely deflated. The LMA is inserted using a single-handed rotational technique. Failed insertion is defined as: failed passage in the pharynx, malposition (air leak) and ineffective ventilation (expired tidal volume<25% of administered volume). The time between picking up the LMA and successful placement is recorded. When failed on the first attempt the LMA will be inserted with a digital guided technique. A Third attempt will be a gum-elastic-bougie guided technique.
3. Oropharyngeal leak pressure is determined at 0-40ml cuff volume in 10 ml increments. The expiratory valve of the circle system is closed at a fixed gas flow of 3 l/min and noting the airway pressure at equilibrium (max allowed 40 cmH2O)
4. Fiber optic position: 4=only vocal cords visible, 3=vocal cords + posterior epiglottis, 2=vocal cords + anterior epiglottis, 1=vocal cords not seen. Fiber optic position will only be evaluated if available at the moment of the study.
5. Cuff pressure is set at 65 cmH2O using a manometer and patients lungs are ventilated at a tidal volume of 10 ml/kg, at a respiratory rate of 12/min. Presence of air leak is detected by listening over the mouth, gastric air leak (stethoscope over epigastrium, larynx, drain tube air leaks (lubricant over proximal end) or end-tidal CO2 > 45 mmHg. Respiratory settings are changed at the discretion of the anesthesiologist after successful placement.
6. Correct gastric tube placement is assessed by suction of fluid. Cardiorespiratory data are collected: bradycardia >100/min, tachycardia >, hypotension, hypoxaemia
7. Upon removal of the LMA at the end of the procedure the device will be checked for blood staining.
8. At discharge from day surgery unit patients will be asked for presence of sore throat.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned for elective minor surgery in the ambulatory surgery unit, who are ASA I or II or III, aged 19-71 years, whose operation is routinely done with a Laryngeal Mask Airway in the supine position.

Exclusion Criteria:

* Patients are excluded if they are <19 or >71 years, have an anticipated difficult airway, a body mass index > 35kg.m-2 or are at risk of aspiration.

Ages: 19 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Airway Leak Pressure | perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ghent, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acx E, Van Caelenberg E, De Baerdemaeker L, Coppens M. Laryngeal mask airway protector generates higher oropharyngeal leak pressures compared to the laryngeal mask airway supreme: A randomized clinical trial in the ambulatory surgery unit. J Anaesthesiol Clin Pharmacol. 2021 Apr-Jun;37(2):221-225. doi: 10.4103/joacp.JOACP_416_19. Epub 2021 Jul 15. PMID 34349370